CLINICAL TRIAL: NCT03978130
Title: REhabilitation at Home uSIng mobiLe Health In oldEr Adults After hospitalizatioN for Ischemic hearT Disease
Acronym: RESILIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-02017
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: partial mask (outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth-CR (Experimental): Participants in this arm will receive the mHealth-CR intervention.
  Interventions: Other: mHealth-CR
- Usual Care (No Intervention): Participants in this arm receive usual care.

INTERVENTIONS:
Other: mHealth-CR — Study participants randomized to the intervention (mHealth-CR) arm during the (in-hospital) baseline visit will receive 3 components for their home activity: (1) communication with exercise therapist (in-hospital assessment/counseling followed by regular communication post-discharge), (2) mHealth-CR software, and (3) wearable activity monitoring device.
  Arms: mHealth-CR

SUMMARY:
RESILIENT is a phase II, multi-center, prospective, pragmatic randomized clinical trial with blinded assessment of the primary endpoint. This study aims to evaluate whether mHealth-CR improves functional capacity in older adults (age ≥65) with IHD compared with standard traditional cardiac rehabilitation care. A total of 400 eligible patients will be randomized in 3:1 manner to mHealth-CR versus usual care for assessment of primary endpoint. Enrollment will occur over approximately 42 months with an expected minimum of 3 months follow-up per participant.

DETAILED DESCRIPTION:
The primary objective of RESILIENT is to evaluate whether mobile health cardiac rehab (mHealth-CR) improves functional capacity in older adults (age ≥65) with ischemic heart disease (IHD), identified at the time of acute myocardial infarction (AMI), percutaneous coronary intervention (PCI), or coronary artery bypass graft (CABG), compared with usual care. Our central hypotheses related to efficacy are that mHealth-CR will (1) improve functional capacity (primary outcome), (2) improve goal attainment, health status, and activities of daily living, and (3) lower rates of hospital readmission and death (secondary outcomes). Our central hypothesis related to engagement is that we will identify distinct trajectories of engagement and characteristics that predict membership in each category.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65
2. Currently hospitalized for AMI, PCI, or CABG or Hospitalized for AMI, PCI or CABG within prior 2 weeks.
3. Capable of self-consent.
4. Understand and are able to perform study procedures (i.e. 6-minute walk test, use mHealth in English or Spanish).

Exclusion Criteria:

1. Non-ambulatory.
2. Moderate or severe cognitive impairment.
3. Unable/unwilling to consent.
4. PCI-related groin hematoma that precludes brisk walking.
5. Incarcerated.
6. Unable to use mHealth software in English or Spanish.
7. Severe osteoarthritis, or joint replacement within last 3 months.
8. Parkinson's disease or other progressive movement disorder.
9. Regular use of walker for ambulation.
10. Projected life expectancy <3 months.
11. Clinical judgment concerning other safety or nonadherence issues.
12. Participants admitted from long-term care facility.
13. Currently listed for heart transplant.
14. Left ventricular assist device recipient.
15. Completion of ambulatory cardiac rehabilitation program within prior 3 months.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Dodson, MD, Principal Investigator — New York Langone Health
Locations (2):
- United States (2):
  - UMass Chan Medical School, Worcester, Massachusetts
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to john.dodson@nyumc.org. To gain access, data requestors will need to sign a data access agreement. The investigator who proposed to use the data.

REFERENCES:
- [Derived] Barua S, Upadhyay D, Pena S, McConnell R, Varghese A, Adhikari S, LeRoy E, Schoenthaler A, Dodson JA. Adherence to Accelerometer Use in Older Adults Undergoing mHealth Cardiac Rehabilitation: Secondary Analysis of a Randomized Clinical Trial. J Med Internet Res. 2025 Dec 23;27:e80522. doi: 10.2196/80522. PMID 41435373
- [Derived] Dodson JA, Adhikari S, Schoenthaler A, Hochman JS, Sweeney G, George B, Marzo K, Jennings LA, Kovell LC, Vorsanger M, Pena S, Meng Y, Varghese A, Johanek C, Rojas M, McConnell R, Whiteson J, Troxel AB. Rehabilitation at Home Using Mobile Health for Older Adults Hospitalized for Ischemic Heart Disease: The RESILIENT Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2453499. doi: 10.1001/jamanetworkopen.2024.53499. PMID 39775808
- [Derived] Dodson JA, Schoenthaler A, Sweeney G, Fonceva A, Pierre A, Whiteson J, George B, Marzo K, Drewes W, Rerisi E, Mathew R, Aljayyousi H, Chaudhry SI, Hajduk AM, Gill TM, Estrin D, Kovell L, Jennings LA, Adhikari S. Rehabilitation Using Mobile Health for Older Adults With Ischemic Heart Disease in the Home Setting (RESILIENT): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Mar 3;11(3):e32163. doi: 10.2196/32163. PMID 35238793

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | mHealth-CR | Usual Care
Started | 298 | 102
Completed | 271 | 85
Not Completed | 27 | 17
Not completed — Lost to Follow-up | 13 | 14
Not completed — Withdrawal by Subject | 12 | 2
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mHealth-CR | Usual Care | Total
Number analyzed (Participants) | 298 | 102 | 400
Age, Continuous [Median (Full Range); unit: years] | 71 [65 to 91] | 71 [65 to 89] | 71 [65 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 27 | 109
  Male | 216 | 75 | 291
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 11 | 34
  Not Hispanic or Latino | 275 | 91 | 366
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 9 | 36
  White | 229 | 74 | 303
  More than one race | 31 | 13 | 44
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 298 | 102 | 400

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walking Distance (6MWD)
Description: Change in 6MWD, reflective of functional capacity, is measured by the 6-minute walk test (6MWT). The 6-minute walk test (6MWT) is a submaximal exercise test in which the pace is self-selected by the participant. The 6MWT will be performed during baseline hospitalization and at the 3-month follow-up visit by a blinded research nurse. The outcome change in 6MWD is calculated as 3 month 6MWD minus baseline 6MWD.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mHealth-CR | Usual Care
Number analyzed (Participants) | 298 | 102
meters | 41.2 (1.5) | 25.6 (2.7)

2. Primary Outcome: Number of Participants in Each Engagement Phenotype on Intervention Arm
Description: Weekly engagement will be measured as the fraction of the following 11 elements completed each week: (1-7) daily entry of exercise data and relative perceived exertion (RPE); (8) completed weekly phone call with exercise therapist; (9) at least one electronic communication with exercise therapist; (10) watching educational video (which will vary by week); and (11) at least one home BP measurement. Engagement will be assessed as a pseudo-continuous outcome, as the score can range from 0% (0 activities completed) to 100% (all 11 activities completed). The participants in the intervention arm will be grouped into 3 engagement phenotypes based on their scores: 1) Persistently Low, 2) Intermediate Declining, and 3) Persistently High.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Persistently Low: Participants who had persistently low engagement.
- Intermediate Declining: Participants who had moderate engagement, but not consistent.
- Persistently High: Participants who had continuously high engagement with the program.
Arm/Group | Persistently Low | Intermediate Declining | Persistently High
Number analyzed (Participants) | 298 | 298 | 298
Participants | 81 | 93 | 124

3. Secondary Outcome: Percentage of Participants With Goal Attainment, as Measured Using a 5-point Goal Attainment Scale (GAS)
Description: Using the SMART goal framework, GAS describes the person's expected level of goal achievement over 3 months, ranging from no change (scored as -2) to much better than expected (scored as +2) out of a 5 point-scale. Scales are dynamically set according to a person's needs, while measurement of attainment is standardized. Overall score is calculated by incorporating the goal of outcomes scores into an aggregated t-score. Goal attainment, through goal setting, is an especially important outcome in older adults who may begin an intervention with a variety of deficits (therefore necessitating individualized therapy towards realistic goals).
Time Frame: 3 months
Measure: Number; unit: Percentage of participants
Arm/Group | mHealth-CR | Usual Care
Number analyzed (Participants) | 298 | 102
Percentage of participants | 25.7 | 20.9

4. Secondary Outcome: 12-Item Short Form Survey (SF-12) Score
Description: The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. For the SF-12, the 3 month score will be analyzed using a threshold of 5 points in SF-12 physical component score (PCS) as a clinically meaningful change.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mHealth-CR | Usual Care
Number analyzed (Participants) | 298 | 102
score on a scale | 46.3 (1) | 48.2 (1.1)

5. Secondary Outcome: Percentage of Participants With no Residual Angina, as Measured by the Seattle Angina Questionnaire 7 (SAQ-7) (Disease-specific Health Status)
Description: The Seattle Angina Questionnaire-7 (SAQ-7) is a self-administered questionnaire that measures patient-reported health measures related to coronary artery disease (CAD). The SAQ-7 is scored from 0 to 100, with higher scores indicating better health status, less frequent angina, and better quality of life (0-24: Poor health status; 25-49: Fair; 50-74: Good; 75-100: Excellent). For SAQ-7, we will analyze at a single time point (3 months) the number of participants who have residual angina (SAQ-7<100) vs. no angina (SAQ-7=100).
Time Frame: Baseline, 3 months
Measure: Number; unit: Percentage of participants
Arm/Group | mHealth-CR | Usual Care
Number analyzed (Participants) | 298 | 102
Percentage of participants | 25.7 | 20.9

6. Secondary Outcome: Percentage of Participants Who Have Any ADL or IADL Impairment
Description: Defined as any improvement or worsening in basic (BADLs) or instrumental (IADLs) over 3 months. The Bristol Activities of Daily Living Scale (BADL) measures basic self-care behaviors: feeding, toileting, bathing, dressing, and ambulating. The score is interpreted based on the total score, which ranges from 0 to 60. Higher scores indicate greater independence in daily living activities. The Lawton Instrumental Activities of Daily Living (IADL) scale measures activities that allow a person to live independently (e.g. food preparation, medication management, transportation, shopping, managing finances, using the telephone, and housekeeping). The total score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
Time Frame: Baseline, 3 months
Measure: Number; unit: percentage of participants
Arm/Group | mHealth-CR | Usual Care
Number analyzed (Participants) | 298 | 102
percentage of participants | 9.7 | 10.6

7. Secondary Outcome: Number of Hospital Readmissions
Description: Defined as number of participants who were readmitted into the hospital with an overnight stay (including observation) in any hospital within 12 months of hospitalization. Data are obtainable via the electronic health record (EHR).
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth-CR | Usual Care
Number analyzed (Participants) | 298 | 102
Participants | 56 | 16

8. Secondary Outcome: Number of Participants Who Died From Any Cause
Description: Data are obtainable via the electronic health record (EHR).
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth-CR | Usual Care
Number analyzed (Participants) | 298 | 102
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed for 3 months. All-Cause Mortality monitored/assessed through follow up, up to 1 year.
Arm/Group | mHealth-CR | Usual Care
All-Cause Mortality (participants affected / at risk) | 5/298 | 1/102
Serious Adverse Events (participants affected / at risk) | 19/298 | 4/102
Other Adverse Events (participants affected / at risk) | 64/298 | 18/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mHealth-CR (N=298) | Usual Care (N=102)
Fall (Musculoskeletal and connective tissue disorders) | 2 | 0
Abnormal labs (Investigations) | 1 | 0
Urinary obstruction (Renal and urinary disorders) | 0 | 1
Planned procedure (Surgical and medical procedures) | 0 | 1
Cancer (Immune system disorders) | 1 | 0
Dizziness (Musculoskeletal and connective tissue disorders) | 1 | 0
COVID (Respiratory, thoracic and mediastinal disorders) | 1 | 0
GI Issues (Gastrointestinal disorders) | 3 | 0
Difficulty Swallowing (Gastrointestinal disorders) | 1 | 0
Chest pain, tightness, angina (Cardiac disorders) | 2 | 0
Planned procedure (Cardiac disorders) | 2 | 1
Heart Failure (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Arrythmia, claudication, hypertensive or hypotensive urgency (Cardiac disorders) | 4 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mHealth-CR (N=298) | Usual Care (N=102)
Cardiac related events (Chest pain, planned procedure, and other) (Cardiac disorders) | 24 | 11
Body pain (Musculoskeletal and connective tissue disorders) | 11 | 3
Fall (Musculoskeletal and connective tissue disorders) | 8 | 1
Other events (Investigations) | 21 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT03978130/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT03978130/ICF_000.pdf